CLINICAL TRIAL: NCT05337384
Title: The Value of Venous Doppler Imaging in Predicting the Indication of Emergency Dialysis in Patients With End-Stage Renal Disease
Brief Title: Sonographic Venous Doppler Imaging in End-Stage Renal Disease
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Mehmet Ali Aslaner, Assoc. Prof., Gazi University
Other Study IDs: GaziU2
Record Dates: First submitted 2022-04-13; First posted 2022-04-20 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Emergent Dialysis; Venous Doppler Ultrasound
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Sonography — Sonographic Venous Doppler Imaging

SUMMARY:
Patients with end-stage renal disease (ESRD) may visit to emergency services for urgent hemodialysis or other reasons. Hemodialysis application in emergency conditions is generally not as optimal as in dialysis units. It takes time to provide suitable conditions (personnel and equipment), the length of stay of patients in the emergency services is prolonged, and this may cause disruption of patient care in these areas where rapid patient care is provided. Therefore, the management of ESRD patients continues to be one of the serious problems faced by emergency physicians.

Sonographic evaluation of the venous system (vena cava inferior, hepatic, portal and renal vein) may be an alternative diagnostic method for need for urgent hemodialysis. Hereby, patients who don't need hemodialysis safely can be discharged from emergency services. Studies conducted so far have generally been based on predicting cardiorenal AKI and renal poor outcomes and have been designed in general ICU conditions.

In this study, the researchers aimed to determine the diagnostic value of sonographic venous Doppler imaging the need for urgent hemodialysis in ESRD patients in the emergency services.

ELIGIBILITY:
Inclusion Criteria:

* Patients with end-stage renal disease

Exclusion Criteria:

* Who are pregnant,
* With cirrhosis and liver malignancy,
* Who do not give consent for the study,
* Arrest presentation
* Unable to scan in the first six hours

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emergency department patients with end-stage renal disease
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
The diagnostic accuracy of sonographic venous Doppler imaging for the need for urgent hemodialysis | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University Faculty of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No